CLINICAL TRIAL: NCT00991289
Title: The Activity of Nitazoxanide in Addition to Peginterferon Alfa-2a and Ribavirin in Chronic Hepatitis C Treatment-Naive Genotype 1 Subjects With HIV Coinfection
Brief Title: Nitazoxanide Plus Ribavirin and Peginterferon for Therapy of Treatment Naive HCV Genotype 1 and HIV Coinfected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5269; 10764 (Registry Identifier: DAIDS ES); ACTG A5269 (Other: ACTG)
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2019-01

CONDITIONS: HIV Infection; Hepatitis C Infection
Keywords: Hepatitis C genotype 1; HCV treatment naive; HCV/HIV coinfection; Antiretroviral; Ribavirin; Pegylated Interferon alfa; Nitazoxanide
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — nitazoxanide; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NTZ/PEG/RBV (Experimental): Participants received nitazoxanide (NTZ) alone for 4 weeks followed by 48 weeks of NTZ with pegylated interferon (PEG) and ribavirin (RBV). Participants who did not achieve early virologic response (EVR) at Week 16 or had detectable hepatitis C virus (HCV) viral load at Week 28 discontinued treatment.
  Interventions: Drug: Nitazoxanide (NTZ); Drug: Pegylated interferon alfa-2a (PEG); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Nitazoxanide (NTZ) — 500 mg twice daily, taken orally with food
  Other Names: Alinia
Drug: Pegylated interferon alfa-2a (PEG) — 180 micrograms via subcutaneous injection once weekly
  Other Names: Pegasys
Drug: Ribavirin (RBV) — Weight-based dosing; 1,000 mg daily, taken orally, for people weighing less than 75 kg or 1,200 mg for people weighing at least 75 kg.
  Other Names: Copegus

SUMMARY:
Infection with hepatitis C virus (HCV) can cause liver scarring, or cirrhosis, and this usually occurs more rapidly among people infected with both HCV and human immunodeficiency virus (HIV). People infected with both HCV and HIV have poor response to the current HCV treatments. This phase II pilot study evaluated whether adding a new HCV medication improves response to the current standard HCV treatment with pegylated interferon and ribavirin in people with both HCV and HIV.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) is a significant cause of liver scarring, or cirrhosis, and accounts for up to 30% of all liver transplants in the United States. People infected with HIV are at a high risk of coinfection with HCV, and the combination of these two infections appears to accelerate progression to cirrhosis. Current treatment for HCV infection includes a 48-week course of two medications taken together, peginterferon alfa-2a (PEG) and ribavirin (RBV). This combination is only effective in 14% to 29% of people infected with both HIV and HCV genotype 1 (the genotype most common in the United States). Further complicating treatment, antiretrovirals (which are used to treat HIV) and HCV medications can often have high toxicity when taken together, limiting dosing.

Nitazoxanide (NTZ) is a medication currently approved to treat intestinal infections that is being investigated for use in treating HCV. NTZ has few side effects and has been shown to increase effectiveness of HCV treatment when combined with PEG and RBV among HCV monoinfected people. This study will test whether adding NTZ to PEG+RBV regimen for people coinfected with HCV and HIV improves HCV treatment outcomes.

Participation in this study will last up to 76 weeks. At study entry, participants completed a brief physical exam, provided a urine sample for a routine safety test, provided a blood sample, and completed a pregnancy test. Participants then initiated NTZ, which they took twice a day with food for up to a year. After 4 weeks on NTZ, participants completed the second study visit, at which they completed the same assessments as at study entry and were asked about the medications they were taking. At this visit, participants initiated the other two study drugs, PEG and RBV. PEG was delivered via injection weekly and RBV was taken orally twice a day with dose dependent on participant's weight at entry.

Participants took NTZ, PEG and RBV together for up to 48 weeks. During this time, participants completed study visits every 4 weeks until Week 52 and then completed follow-up visits at Weeks 64 and 76. At these visits, participants completed the same assessments as at previous visits, and, at certain weeks, also fasted for 8 hours before blood draw. Additional blood samples were collected and stored at Weeks 4, 8, 16, 52 and 76 in order to do future testing.

Participants who did not achieve an early virologic response to the study treatment (at least a 2-log10 decrease in HCV viral load or undetectable HCV viral load at Week 16), or had detectable HCV viral load at Week 28), stopped study treatment and discontinued study early, at about 20 or 32 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Documentation of hepatitis C virus (HCV) genotype 1 infection prior to entry
* Chronic HCV infection for at least 180 days
* CD4+ cell count greater than 200 cells/mm3 obtained within 90 days prior to study entry
* Detectable HCV viral load obtained within 90 days prior to study entry
* Any change in antiretroviral (ARV) regimen, including initiation of antiretroviral therapy (ART), a switch in ART regimen, or a discontinuation of ART, had to have occurred more than 60 days prior to study entry. Breaks in therapy for a maximum of 14 days total during the 60-day period were allowed. Participants not on ART should have had no plans to initiate therapy during the first 24 weeks after study entry. Participants who did start ART did not have to discontinue study treatment. Participants on ART should have planned to remain on the same therapy for at least 12 weeks after study entry. Changes in formulation or dosage were permitted.
* Certain laboratory values obtained within 42 days prior to study entry
* Agreement to use contraception, if participating in sexual activity that could lead to pregnancy, for the duration of study and for 6 months afterward
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase less than or equal to five times the upper limit of normal (ULN)
* Hemoglobin >=11 g/dl for men and >=10 g/dl for women

Exclusion Criteria:

* Use of the ARV didanosine (ddI)
* Receipt of any interferon
* Receipt of any therapy for HCV, including ribavirin (RBV) or experimental treatment
* Decompensated cirrhosis
* Currently active or other known causes of significant liver disease, including chronic or acute hepatitis B, acute hepatitis A, hemochromatosis, or homozygous alpha-1 antitrypsin deficiency
* Pregnancy or breastfeeding
* Men with pregnant sexual partners or men planning pregnancy with any sexual partner during treatment or for 24 weeks after treatment completion
* Uncontrolled or active depression, other psychiatric disorder, or any hospitalization within the past 52 weeks that, in the opinion of the site investigator, would prevent participation
* Prior suicide attempt
* Active thyroid disease (use of thyroid hormone replacement therapy permitted if thyroid stimulating hormone [TSH] or free thyroxine [T4] in the normal range)
* History of autoimmune processes, including Crohn's disease, ulcerative colitis, severe psoriasis, or rheumatoid arthritis, that may be exacerbated by interferon use
* Systemic antineoplastic or immunomodulatory treatment or radiation within 24 weeks prior to study entry
* Serious illness, including malignancy or active coronary artery disease, within 24 weeks prior to study entry
* Chronic medical condition that, in the site investigator's opinion, might preclude completion of the protocol
* Presence of acute or active opportunistic infections within 24 weeks prior to study entry
* Evidence of hepatocellular carcinoma (HCC) or alpha-fetoprotein level of greater than 50 ng/ml unless an imaging procedure (e.g., computed tomography [CT] scan or magnetic resonance imaging [MRI]) showed no evidence of a hepatic tumor. Each may have been obtained up to 24 weeks before study entry.
* History of hemoglobinopathy (e.g., thalassemia) or any other cause of or tendency toward hemolysis
* History of major organ transplantation with an existing functional graft
* Known allergy, sensitivity, or any hypersensitivity to components of study drugs or their formulations
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Peters, MD, Study Chair — University of California, San Francisco
Locations (18):
- United States (17):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Rossignol JF, Elfert A, El-Gohary Y, Keeffe EB. Improved virologic response in chronic hepatitis C genotype 4 treated with nitazoxanide, peginterferon, and ribavirin. Gastroenterology. 2009 Mar;136(3):856-62. doi: 10.1053/j.gastro.2008.11.037. Epub 2008 Nov 19. PMID 19135998
- [Background] Korba BE, Montero AB, Farrar K, Gaye K, Mukerjee S, Ayers MS, Rossignol JF. Nitazoxanide, tizoxanide and other thiazolides are potent inhibitors of hepatitis B virus and hepatitis C virus replication. Antiviral Res. 2008 Jan;77(1):56-63. doi: 10.1016/j.antiviral.2007.08.005. Epub 2007 Sep 4. PMID 17888524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women at least 18 years of age with genotype 1 hepatitis C virus (HCV) and human immunodeficiency virus (HIV) coinfection and naive to previous HCV treatment were recruited for participation in this study.
Groups:
- NTZ/PEG/RBV: Participants received nitazoxanide (NTZ) alone for 4 weeks followed by up to 48 weeks of NTZ with pegylated interferon (PEG) and ribavirin (RBV). Participants who did not achieve early virologic response (EVR) at Week 16 or had detectable hepatitis C virus (HCV) viral load at Week 28 discontinued treatment.
Period: Overall Study
Arm/Group | NTZ/PEG/RBV
Started | 67 (68 participants enrolled, one was found to have been ineligible and was excluded.)
COMPLETED Week 16 | 61 (Completed 16 weeks of the study (the primary endpoint time point). The study continued to Week 76.)
Completed | 55 (Completed study.)
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (8.5)
Age, Customized [Number; unit: participants]
  <25 years | 1
  25 to <30 years | 1
  30 to <35 years | 4
  35 to <40 years | 3
  40 to <45 years | 11
  45 to <50 years | 13
  50 to <55 years | 18
  55 to 60 years | 13
  >=60 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 52
Race/Ethnicity, Customized [Number; unit: Participants] — Race/ethnicity, self-reported (NIH categories)
  Participants
    White, Non-Hispanic | 21
    Black, Non-Hispanic | 32
    Hispanic, Regardless of Race | 12
    Other/Unknown | 2
Region of Enrollment [Number; unit: participants]
  United States | 67
HCV viral load level [Median (Inter-Quartile Range); unit: log10 IU/ml] — Hepatitis C virus (HCV) viral load testing was done using Cobas AmpliPrep/Taqman HCV Test with lower limit of quantitation of 43 IU/ml.
  log10 IU/ml | 6.4 [6.0 to 6.7]
CD4+ T cell count [Median (Inter-Quartile Range); unit: cells/mm3] | 452 [323 to 738]
Number of participants with indicated HIV viral load [Number; unit: participants] — A blood sample was drawn to determine the HIV viral load by local laboratories. HIV viral load was categorized as <lower limit of quantification (undetectable) of the assay or >=lower limit of quantification of the assay (detectable). The assays used were bDNA assay (Versant HIV-1 RNA 3.0), Roche COBAS AmpliPrp/Taqman HIV-1 assay and Abbott RealTime HIV-1 assay.
  participants
    Undetectable HIV viral load | 49
    Detectable HIV viral load | 16
    Unknown | 2
HIV Antiretroviral therapy (ART) status [Number; unit: participant]
  On ART | 61
  Not on ART | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: Complete early virologic response (cEVR) was defined as undetectable HCV viral load (<43 IU/ml) at week 16, where 43 is the lower limit of quantification of the assay (Cobas AmpliPrep/Taqman HCV Test).
Time Frame: Week 16
Population: All participants who enrolled, except one participant who was found to have been ineligible after entry. The analysis was intention to treat wherein participants who dropped out early without Week 16 HCV viral load result were considered non-responders.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
percentage of participants | 38.8 [28.8 to 49.6]

2. Primary Outcome: Percentage of Participants With Early Virologic Response (EVR)
Description: Early virologic response (EVR) was defined as undetectable HCV viral load (<43 IU/ml) at Week 16 or at least a 2-log10 decrease in HCV viral load from study entry at Week 16, where 43 is the lower limit of quantification of the assay (Cobas AmpliPrep/Taqman HCV Test).
Time Frame: Weeks 0, 16
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
percentage of participants | 65.7 [55.0 to 75.3]

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR)
Description: Sustained virologic response (SVR) was defined as undetectable HCV viral load (<43 IU/ml) at 24 weeks after treatment discontinuation, where 43 is the lower limit of quantification of the assay (Cobas AmpliPrep/Taqman HCV Test). Participants who failed to achieve EVR or had detectable HCV RNA at Week 28 and per protocol discontinued study, and participants without HCV RNA from 24 weeks after treatment discontinuation, were considered non-responders.
Time Frame: 24 weeks after treatment discontinuation
Population: All participants who enrolled, except one who was found to have been ineligible after entry. The analysis was intention to treat wherein participants who dropped out early without HCV RNA from 24 weeks after treatment discontinuation, non-EVRs and those with detectable HCV RNA at Week 28, were considered non-responders.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
percentage of participants | 32.8 [23.4 to 43.5]

4. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR)
Description: Rapid virologic response (RVR) was defined as undetectable HCV viral load (<43 IU/ml) at Week 8 where 43 is the lower limit of quantification of the assay (Cobas AmpliPrep/Taqman HCV Test).
Time Frame: Week 8
Population: All participants who enrolled, except one participant who was found to have been ineligible after entry. The analysis was intention to treat wherein participants who dropped out early without Week 8 HCV viral load result were considered non-responders.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
percentage of participants | 10.4 [5.0 to 18.7]

5. Secondary Outcome: Number of Participants With Adverse Events of Grade 2 or Higher
Description: Number of participants who experienced an adverse event of Grade 2 or higher at any time after study entry. Grading of adverse events (signs and symptoms and laboratory toxicities) was according to Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004.
Time Frame: From study entry to up to week 76
Population: All participants who enrolled, except one participant who was found to have been ineligible after entry.
Measure: Number; unit: participants
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
participants | 65

6. Secondary Outcome: Change in Hemoglobin Level From Study Entry
Description: Change in hemoglobin (HGB) was calculated as HGB at later time point (Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 76) minus HGB at study entry.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 76.
Population: All participants who enrolled (except one participant who was found to have been ineligible after entry) and had HGB measurements available at entry and at the respective post-entry time point.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
g/dL
  Change in HGB at Week 4: number analyzed (Participants) | 65
  Change in HGB at Week 4 | -0.1 [-0.6 to 0.4]
  Change in HGB at Week 8: number analyzed (Participants) | 65
  Change in HGB at Week 8 | -2.1 [-3.0 to -1.1]
  Change in HGB at Week 12: number analyzed (Participants) | 63
  Change in HGB at Week 12 | -2.5 [-3.5 to -1.8]
  Change in HGB at Week 16: number analyzed (Participants) | 60
  Change in HGB at Week 16 | -2.5 [-3.5 to -1.4]
  Change in HGB at Week 20: number analyzed (Participants) | 55
  Change in HGB at Week 20 | -2.5 [-3.8 to -1.3]
  Change in HGB at Week 24: number analyzed (Participants) | 51
  Change in HGB at Week 24 | -2.4 [-3.2 to -1.3]
  Change in HGB at Week 28: number analyzed (Participants) | 45
  Change in HGB at Week 28 | -2.5 [-3.4 to -1.6]
  Change in HGB at Week 32: number analyzed (Participants) | 38
  Change in HGB at Week 32 | -2.7 [-3.4 to -1.7]
  Change in HGB at Week 36: number analyzed (Participants) | 39
  Change in HGB at Week 36 | -2.5 [-3.9 to -1.7]
  Change in HGB at Week 40: number analyzed (Participants) | 40
  Change in HGB at Week 40 | -2.6 [-3.4 to -2.1]
  Change in HGB at Week 44: number analyzed (Participants) | 31
  Change in HGB at Week 44 | -2.6 [-3.9 to -1.6]
  Change in HGB at Week 48: number analyzed (Participants) | 32
  Change in HGB at Week 48 | -2.7 [-3.4 to -1.9]
  Change in HGB at Week 52: number analyzed (Participants) | 31
  Change in HGB at Week 52 | -2.9 [-3.8 to -1.6]
  Change in HGB at Week 76: number analyzed (Participants) | 29
  Change in HGB at Week 76 | -0.9 [-1.3 to -0.5]

7. Secondary Outcome: Percent Change in Fasting Insulin Level From Study Entry
Description: Percent Change in fasting insulin (FINS) was calculated as FINS at later time point (16, 28, 52, 76) minus FINS at study entry, divided by FINS at study entry x 100%. Study protocol required fasting for at least 8 hours (nothing by mouth except medications and water) prior to specimen collection for fasting insulin testing.
Time Frame: Weeks 0, 16, 28, 52, and 76
Population: All participants who enrolled (except one participant who was found to have been ineligible after entry) and had FINS measurements available at entry and the respective post-entry time point.
Measure: Median (Inter-Quartile Range); unit: percentage of FINS at study entry
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
percentage of FINS at study entry
  Percent change in FINS at Week 16: number analyzed (Participants) | 58
  Percent change in FINS at Week 16 | 0 [-30.8 to 64.7]
  Percent change in FINS at Week 28: number analyzed (Participants) | 40
  Percent change in FINS at Week 28 | 8.8 [-33.2 to 67.9]
  Percent change in FINS at Week 52: number analyzed (Participants) | 28
  Percent change in FINS at Week 52 | 28.2 [-15.0 to 87.5]
  Percent change in FINS at Week 76: number analyzed (Participants) | 23
  Percent change in FINS at Week 76 | 8.3 [-48.0 to 56.3]

8. Secondary Outcome: Percent Change in Fasting Glucose Level From Study Entry
Description: Percent Change in fasting glucose (FGLUC) was calculated as FGLUC at later time point (16, 28, 52, 76) minus FGLUC at study entry, divided by FGLUC at study entry x 100%. Study protocol required fasting for at least 8 hours (nothing by mouth except medications and water) prior to specimen collection for fasting glucose testing.
Time Frame: Weeks 0, 16, 28, 52, and 76
Population: All participants who enrolled (except one participant who was found to have been ineligible after entry) and had FGLUC measurements available at entry and the respective post-entry time point.
Measure: Median (Inter-Quartile Range); unit: percentage of FGLUC at study entry
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
percentage of FGLUC at study entry
  Percent change in FGLUC at Week 16: number analyzed (Participants) | 58
  Percent change in FGLUC at Week 16 | -3.2 [-12.6 to 7.0]
  Percent change in FGLUC at Week 28: number analyzed (Participants) | 41
  Percent change in FGLUC at Week 28 | -5.3 [-9.9 to 4.9]
  Percent change in FGLUC at Week 52: number analyzed (Participants) | 29
  Percent change in FGLUC at Week 52 | 1.1 [-11.8 to 8.0]
  Percent change in FGLUC at Week 76: number analyzed (Participants) | 24
  Percent change in FGLUC at Week 76 | 0 [-7.4 to 8.4]

9. Secondary Outcome: Percent Change in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) From Study Entry
Description: HOMA-IR was calculated as [fasting glucose (mg/dL) x fasting insulin (uIU/mL)]/405. Percent Change in HOMA-IR was calculated as HOMA-IR at later time point (16, 28, 52, 76) minus HOMA-IR at study entry, divided by HOMA-IR at study entry x 100%. Study protocol required fasting for at least 8 hours (nothing by mouth except medications and water) prior to specimen collection for fasting insulin and fasting glucose testing.
Time Frame: Weeks 0, 16, 28, 52, and 76
Population: All participants who enrolled (except one participant who was found to have been ineligible after entry) and had fasting insulin and fasting glucose measurements available at entry and the respective post-entry time point.
Measure: Median (Inter-Quartile Range); unit: percentage of HOMA-IR at study entry
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
percentage of HOMA-IR at study entry
  Percent change in HOMA-IR at Week 16 (n=56): number analyzed (Participants) | 56
  Percent change in HOMA-IR at Week 16 (n=56) | -13.0 [-31.6 to 64.2]
  Percent change in HOMA-IR at Week 28 (n=39): number analyzed (Participants) | 39
  Percent change in HOMA-IR at Week 28 (n=39) | -6.3 [-42.7 to 81.1]
  Percent change in HOMA-IR at Week 52 (n=27): number analyzed (Participants) | 27
  Percent change in HOMA-IR at Week 52 (n=27) | 23.2 [-24.2 to 87.1]
  Percent change in HOMA-IR at Week 76 (n=22): number analyzed (Participants) | 22
  Percent change in HOMA-IR at Week 76 (n=22) | 9.5 [-48.0 to 59.5]

10. Secondary Outcome: Change in log10 HCV Viral Load After 4 Weeks of Nitazoxanide (NTZ) Monotherapy.
Description: Change in log10 HCV viral load was calculated as log10-transformed HCV viral load at Week 4 minus log10-transformed HCV viral load at study entry. HCV viral load testing was done using Cobas AmpliPrep/Taqman HCV Test.
Time Frame: Weeks 0, 4
Population: All participants who enrolled, except one participant who was found to have been ineligible after entry, and had HCV viral load measurements available at entry and at Week 4 were analyzed.
Measure: Median (Inter-Quartile Range); unit: log10 IU/mL
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 64
log10 IU/mL | -0.12 [-0.30 to 0.13]

11. Secondary Outcome: Number of Participants With HCV Genotype 1
Description: Confirmatory HCV genotyping was performed on stored plasma from entry using VERSANT HCV Genotype assay v2.0 (LiPA, RUO, Siemens Healthcare Diagnostics Inc., Tarrytown, NY).
Time Frame: Week 0
Population: All participants who enrolled, except one participant who was found to have been ineligible after entry.
Measure: Number; unit: participants
Arm/Group | NTZ/PEG/RBV
Number analyzed (Participants) | 67
participants | 67

ADVERSE EVENTS:
Time Frame: From study entry to Week 76.
Arm/Group | NTZ/PEG/RBV
Serious Adverse Events (participants affected / at risk) | 13/67
Other Adverse Events (participants affected / at risk) | 67/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NTZ/PEG/RBV (N=67)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Syncope (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NTZ/PEG/RBV (N=67)
Anaemia (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 18
Dysphagia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 23
Irritability (General disorders) | 4
Pain (General disorders) | 5
Pyrexia (General disorders) | 5
Pneumonia bacterial (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 36
Aspartate aminotransferase increased (Investigations) | 29
Blood albumin abnormal (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 6
Blood bicarbonate abnormal (Investigations) | 5
Blood bilirubin increased (Investigations) | 14
Blood glucose abnormal (Investigations) | 11
Blood glucose increased (Investigations) | 6
Blood phosphorus decreased (Investigations) | 14
Blood potassium decreased (Investigations) | 6
Blood sodium decreased (Investigations) | 9
Blood triglycerides abnormal (Investigations) | 4
Blood uric acid increased (Investigations) | 11
Haemoglobin decreased (Investigations) | 24
Lipase increased (Investigations) | 11
Neutrophil count decreased (Investigations) | 54
Platelet count decreased (Investigations) | 35
Weight decreased (Investigations) | 21
White blood cell count decreased (Investigations) | 23
Decreased appetite (Metabolism and nutrition disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights